CLINICAL TRIAL: NCT02773628
Title: Impact of Reduction of Dust Mite Allergenic Load on Step Down of Inhaled Corticosteroids in Stable Asthma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: methodological concerns about study design
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK/15-12-127/4581
Record Dates: First submitted 2016-04-25; First posted 2016-05-16 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Placebo Comparator): stable asthmatics receiving an Acar'up placebo system
  Interventions: Device: Acar'up placebo system
- treatment group (Active Comparator): stable asthmatics receiving Acar'up system
  Interventions: Device: Acar'up system

INTERVENTIONS:
Device: Acar'up system
  Arms: treatment group
Device: Acar'up placebo system
  Arms: control group

SUMMARY:
Eviction methods for dust mite allergy have been evaluated in asthma control in a recent Cochrane meta-analysis. None have shown efficacy on asthma control and there are not recommended. The purpose is to evaluate the efficacy of a new commercialized system (Acar'Up) to decrease dust mite load and to assess its impact on the possibility to perform inhaled corticosteroids step down in stable asthmatics.

DETAILED DESCRIPTION:
Eviction methods for dust mite allergy have been evaluated in asthma control in a recent Cochrane meta-analysis. None have shown efficacy on asthma control and there are not recommended. The purpose is to evaluate the efficacy of a new commercialized system, Acar'Up (a spray pulverized on a technical textile that traps the dust mite) to decrease dust mite load and to assess its impact on the possibility to perform inhaled corticosteroids step down in stable asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* confirmed asthma diagnosis
* controlled asthma for more than 3 months
* treatment with inhaled corticosteroids
* dust mite allergy proved by skin tests ou specific immunoglobulin E

Exclusion Criteria:

* chronic obstructive pulmonary disease, bronchiectasis, Fibrosis, tuberculosis
* asthma-chronic obstructive pulmonary disease overlap syndrome
* ongoing desensitization for dust mite
* pregnancy
* previous use of Acar'up

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
assessment of successful stepdown of inhaled corticosteroid using clinical evaluation | 4 months
  assessment of the successful step down of inhaled corticosteroid using clinical evaluation
assessment of successful stepdown of inhaled corticosteroid using asthma scale: asthma control questionnaire (ACQ) | 4 months
  assessment of the successful step down of inhaled corticosteroid using asthma scale: asthma control questionnaire (ACQ)
assessment of successful stepdown of inhaled corticosteroid using asthma quality of life questionnaire (AQLQ) | 4 months
  assessment of the successful step down of inhaled corticosteroid using asthma quality of life questionnaire (AQLQ)

SECONDARY OUTCOMES:
assessment of asthma control by the asthma control questionnaire questionnaire | 4 months
  by the asthma control questionnaire
assessment of asthma quality of life by the asthma quality of life questionnaire | 4 months
  by the asthma quality of life questionnaire
assessment of rhinitis control by the rhinitis quality of life questionnaire | 4 months
  by the rhinitis quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHu Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No